CLINICAL TRIAL: NCT07197879
Title: Effect of Dynamic Sitting on Pain Development - Part 2 - a Randomized Controlled Cross-over Study
Brief Title: Effect of Dynamic Sitting on Pain Development - Part 2
Acronym: DynSit-Pain 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences for Health Professions Upper Austria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2025-05-12
Record Dates: First submitted 2025-09-26; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study Track 1: Group A (Experimental): The pre-existing static office chair will be used in the personal workplace for the first 6 weeks within the first half of the study. A wash-out period of a minimum of 4 weeks will be executed after the first half of the study. A dynamic office chair (saddle chair with standard pendulum mechanism) will be used on the personal workstation for 6 weeks within the second half of the study after the wash-out period.
  Interventions: Device: Dynamic office chair (saddle chair with standard pendulum mechanism)
- Study Track 1: Group B (Experimental): A dynamic office chair (saddle chair with standard pendulum mechanism) will be used in the personal workplace for the first 6 weeks within the first half of the study. A wash-out period of a minimum of 4 weeks will be executed after the first half of the study. The pre-existing static office chair will be used on the personal workstation for 6 weeks within the second half of the study after the wash-out period.
  Interventions: Device: Dynamic office chair (saddle chair with standard pendulum mechanism)
- Study Track 2: Group C (Experimental): The pre-existing static office chair will be used in the personal workplace for the first 6 weeks within the first half of the study. A wash-out period of a minimum of 4 weeks will be executed after the first half of the study. A dynamic office chair (office swivel chair with integrated newly developed pendulum mechanism) will be used on the personal workstation for 6 weeks within the second half of the study after the wash-out period.
  Interventions: Device: Dynamic Office Chair (office swivel chair with integrated newly developed pendulum mechanism)
- Study Track 2: Group D (Experimental): A dynamic office chair (office swivel chair with integrated newly developed pendulum mechanism) will be used in the personal workplace for the first 6 weeks within the first half of the study. A wash-out period of a minimum of 4 weeks will be executed after the first half of the study. The pre-existing static office chair will be used on the personal workstation for 6 weeks within the second half of the study after the wash-out period.
  Interventions: Device: Dynamic Office Chair (office swivel chair with integrated newly developed pendulum mechanism)

INTERVENTIONS:
Device: Dynamic office chair (saddle chair with standard pendulum mechanism) — The dynamic office chair has a typical office chair design (e.g. seat pan and a lumbar support). The seat pan is mounted on a flexible mechanic construction that allows hip movements in the frontal plane while sitting.
  Arms: Study Track 1: Group A; Study Track 1: Group B
Device: Dynamic Office Chair (office swivel chair with integrated newly developed pendulum mechanism) — The dynamic office chair has a typical office chair design (e.g. seat pan and a lumbar support). The seat pan is mounted on a flexible mechanic construction that allows hip movements in the frontal plane while sitting.
  Arms: Study Track 2: Group C; Study Track 2: Group D

SUMMARY:
As a follow-up project to the Dyn-Sit-Pain study, this research aims to investigate the overall health as well as the physical and mental well-being through dynamic office chairs. The development of an innovative dynamic office chair concept will be professionally and scientifically supported, and the developed prototypes will be examined within the framework of usability studies.

DETAILED DESCRIPTION:
This clinical trial is a prospective, randomised, controlled, open-label study with two tracks, each in a cross-over design investigating the effect of of two dynamic office chairs (saddle chair with standard pendulum mechanism [Smart Moving Technology], study track 2 = office swivel chair with integrated newly developed pendulum mechanism [Smart Moving Technology New]) on the musculoskeletal system of office workers classified as pain developers.

The study consists of a pre-screening visit and 4 assessment days / visits. After proving eligibility for the study (inclusion/exclusion criteria), subjects are assigned to one of the two study tracks. Subjects are randomised to one of the two study tracks and then to the respective group (Group A to D).

* Study track 1: saddle chair with standard pendulum mechanism (= intervention 1) + static office chair (= control)
* Study track 2: office swivel chair with integrated newly developed pendulum mechanism (= intervention 2) + static office chair (= control).

Depending on the study track and group allocation, the test subjects first receive a dynamic office chair (= intervention) or a static office chair (= control). The randomization will be realized with opaque envelopes in different colours and follows international recommendations.

Overall participants will execute identical assessments. A wash-put period between the control and the intervention phases ensures identical baseline conditions. The overall duration of study participation equals 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed consent
* People aged between 18 and 65 years
* People classified as pain developers (e.g.: a 10 mm increase in pain on a 100 mm paper-based VAS)
* Office workers
* Employment status: > 25 h / week
* Sufficient knowledge of German (min. B2 level)
* Body height of at least 160cm required
* Electrically or manually height-adjustable table at main workstation

Exclusion Criteria:

* Physical or mental limitations that make dynamic sitting or use of the procedure chair difficult (e.g. wheelchair users, vestibular dysfunction)
* Pregnancy
* Sitting for less than 20 hours per week at the main workplace
* Body weight over 110 kg and a body height over 195 cm
* Regular therapy or medication for pain or medication that affects the perception of pain (e.g. certain psychotropic drugs according to the package leaflet)
* office chair to which it is not possible to attach the swivel mechanism prototype
* Presence of any chronic disease that may influence pain perception (e.g., chronic kidney disease, fibromyalgia, neuropathy, chronic fatigue syndrome)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in subjective lower back pain (before vs. after work, weekly average) estimated by visual analogue scale (VAS) | 6 weeks
  Participants will rate their subjectively perceived lower back pain before and after a conventional occupational day on 5 consecutive days starting at baseline (week 1) and ending with the post-intervention visit (week 6). Subjectively perceived lower back pain will be assessed with a Visual Analogue Scale (VAS). The VAS used for this study ranges from 0 (none) to 100 points (strongest pain imaginable).
  Question: Please rate the level of your lower back pain at this moment.

SECONDARY OUTCOMES:
Mean change in subjective mental fatigue (before vs. after work, weekly average) estimated by VAS | 6 weeks
  Participants will rate their subjectively perceived mental fatigue before and after a conventional occupational day on 5 consecutive days starting at baseline (week 1) and ending with the post-intervention visit (week 6). Subjectively perceived mental fatigue will be assessed with a Visual Analogue Scale (VAS). The VAS used for this study ranges from 0 (none) to 100 points (strongest mental fatigue imaginable).
  Question: Please rate the level of your mental fatigue at this moment.
Mean subjectively rated work performance (after work, weekly average) estimated by VAS | 6 weeks
  Participants will rate their subjectively perceived working performance before and after a conventional occupational day on 5 consecutive days starting at baseline (week 1) and ending with the post-intervention visit (week 6). Subjectively perceived working performance will be assessed with a Visual Analogue Scale (VAS). The VAS used for this study ranges from 0 (not productive at all) to 100 points (very productive).
  Question: Please rate the level of your working performance on this working day.
Change in impact of pain on the daily life (pre vs. post intervention) estimated by ODI-D | 6 weeks
  Participants will rate their subjectively perceived pain with the German version of the Oswestry Disability Index (ODI-D) at the baseline and post-intervention visits.
  The ODI-D coverts 10 items: Pain intensity, Personal care, Lifting, Walking, Sitting, Standing, Sleeping, Sex (if applicable), Social and Travel. Each item consists of 6 statements which are scored from 0 (lowest disability) to 5 (highest disability).
Usability estimated using the UEQS questionnaire | 6 weeks
  Subjects will rate the usability of the dynamic chair with the German version of the User Experience Questionnaire-Short version (UEQ-S) at the relevant post-intervention visit.
  The UEQ-S cover both classical usability aspects (efficiency, perspicuity, dependability) and user experience aspects (originality, stimulation). It consists of 8 items, each rated on a seven-point scale with a ranked order. The endpoints of the items are (left to right): obstructive to supportive / complicated to easy / inefficient to efficient / confusing to clear / boring to exciting / not interesting to interesting / conventional to inventive and usual to leading edge.
Sitting behaviors estimated by microcontrollers | 6 weeks
  The usage of the interventional chair will be tracked (i.e., the system cannot detect which person is sitting on it) by means of a microcontroller to determine if the dynamic chair was used or replaced within the interventional period.
Number of adverse events estimated from an AEs form sheet | 16 weeks
  In the diary and at all study visits participants will be asked for new adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Applied Sciences for Health Professions Upper Austria, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No